CLINICAL TRIAL: NCT03346447
Title: Effect of Baby Wipe Solutions on Fecal Enzyme-induced Irritation
Status: Completed | Type: Observational
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 500-17-06
Record Dates: First submitted 2017-09-12; First posted 2017-11-17 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Skin Health

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Artificial Fecal Enzyme — Artificial Fecal enzyme Trypsin/Chymotrypsin mixture

SUMMARY:
This is a single-center, prospective, single-blind pilot study to determine baby wipe formulations on an adult dermatitis model.

DETAILED DESCRIPTION:
This is a single-center, prospective, single-blind pilot study to determine baby wipe formulations on an adult dermatitis model.

Biophysical measurements will be taken at each test sites.

ELIGIBILITY:
Inclusion Criteria:

* 1. Fluent in English, willing and able to read, understand, and sign the informed consent form (ICF) 2. Ability to complete the course of the study and comply with instructions; 3. Females aged 18 to 40 years, in good general health as deemed by the investigator (no physical required).

  4. Caucasian individuals with Fitzpatrick skin type I, II, or III (See Appendix I).

  5. Individuals free of any systemic or dermatological disorder including a known history of allergies or other medical conditions which, in the opinion of the investigator, could interfere with the conduct of the study, interpretation of results, or increase the risk of adverse reactions.

  6. Anticipated ability to complete the course of the study and to comply with instructions.

  7. Females practicing an acceptable method of birth control (abstinence is acceptable). Females of child-bearing potential must have practiced an acceptable method of birth control for the past 3 months and be willing to continue using the same method throughout the duration of the study. Acceptable methods of birth control, include: 1) Systemic birth control (Subjects must have been taking the same type of birth control for at least 3 months prior to entering the study and must not change the type of birth control during the study); 2) Condom with spermicide; 3) IUD; 4) Vasectomized partner; and 5) Abstinence. Females who are post-menopausal (for at least 1 year) or have had a permanent sterilization procedure (i.e. hysterectomy, tubal ligation, bilateral oophorectomy) do not need to have additional birth control methods.

Exclusion Criteria:

* 1. Individuals with any visible skin disease, skin condition (e.g., back acne) including baseline erythema assessment > 0.5, or tattoos in the test area (mid to upper back).

  2. Individuals with abnormal skin pigmentation at the test sites, which might interfere with subsequent evaluations of dermal responsiveness.

  3. Individuals with recent prolonged sun or tanning bed exposure in the test area 4. Individuals with excessive dryness or redness at the sites of application. 5. Individuals with a known hypersensitivity to any of the components of the insult, controls, or adhesive tapes.

  6. Subjects must not have applied any lotions, creams, powders, or oils to their backs the morning of the study. Additionally, two hours must have passed since bathing or showering.

  7. Women who are pregnant or nursing. 8. Individuals who have participated on a study involving the test sites (back) in the previous 30 days.

  9. Individuals participating in another clinical study 10. Individuals with open or healing cuts/incisions, abrasions, lesions, pustules, fissures, or broken mucosa/skin in the test area

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of 24 Caucasian females, age 18-40, in good general health and free from dermatological conditions in the testing area.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Erythema | 1 week
  Time for a test site to reach an erythema score of ≥ 2.
Transepidermal Water Loss (TEWL) | 1 week
  difference in TEWL between test sites
pH | 1 week
  difference in pH between test sites
Chromameter redness | 1 week
  difference in redness between test sites

SECONDARY OUTCOMES:
Biophysical Measurement changes of skin capacitance | 1 week
  difference in capacitance between test sites
Microbiome profile | 1 day
  OTUs of microbiome in test site samples

CONTACTS AND LOCATIONS:
Overall Officials: Barry Reece, Principal Investigator — RCTs
Locations (1):
- Reliance Clinical Testing Services, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Subjects will be identified on CRFs and other documents submitted to the Sponsor by their unique identification number with or without their initials, not by name. Documents that identify the subject (e.g., the signed informed consent) are not to be submitted to the Sponsor and must be maintained in confidence by the Investigator.